CLINICAL TRIAL: NCT01825681
Title: Life Enhancing Activities for Family Caregivers (LEAF)
Brief Title: Life Enhancing Activities for Family Caregivers
Acronym: LEAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Glenna Dowling, Professor and chair, Department of Physiological Nursing, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14-13236; A115168 (Other Grant/Funding Number: Atlantic Philanthropies)
Record Dates: First submitted 2013-03-25; First posted 2013-04-08 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Stress; Dementia; Affect
Keywords: positive affect; caregivers; caregiving; stress; mood; dementia; Alzheimer's; FTD; Lewy; mindfulness; help
MeSH Terms: conditions — Dementia; Helping Behavior | interventions — Caregivers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- positive affect intervention (Experimental): positive affect intervention
  Interventions: Behavioral: Positive Affect
- wait list control (No Intervention): wait list control

INTERVENTIONS:
Behavioral: Positive Affect — Six-session skill-building program designed to raise levels of positive emotion when skills are practiced over the duration of the program.
  Other Names: Life Enhancing Activities for Family Caregivers (LEAF)
  Arms: positive affect intervention

SUMMARY:
Life Enhancing Activities for Family Caregivers is a six-week program designed to increase positive affect in people who care for a family member with dementia. The intervention consists of 6 weekly one-hour sessions conducted one-on-one with a trained facilitator to teach simple skills that are practiced at home in a study-supplied workbook. The program is preceded and followed by a 30-45 minute questionnaire. Follow-up assessments will be conducted at 1-month, 3-months, and 6-months post intervention.

Primary hypothesis is that experimental subjects who participate in LEAF will demonstrate significantly greater improvements in psychological outcomes and will engage in more problem focused and positive appraisal forms of coping compared to the wait-list control condition.

DETAILED DESCRIPTION:
All study activities can be conducted from the participant's home, making participation possible for any qualified caregiver with computer and wifi access, in any U.S. state. The LEAF study will supply the tablet computer, software, and workbook required for participation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to be defined as the primary care provider for a family member with dementia. (Person with dementia must live with the caregiver or in their own home and not in a care facility.)
* Must speak and read English
* Must have the ability to provide informed consent

Exclusion Criteria:

* Lack of access to a high speed internet connection
* Evidence of severe cognitive impairment or active psychosis, as assessed by trained interviewers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-10; Primary Completion 2017-08 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Repeated measures of the modified version of the Differential Emotions Scale (DES) (Izard, 1977) | Baseline and weeks 6 and 10; 3-months and 6-months post
  The DES will be used to assess positive and negative affect. This 20-item version of the DES was modified to include additional positive affect items as well as those that are likely to tap into trait positive affectivity. The full scale assesses interest, enjoyment, surprise, sadness, anger, disgust, contempt, fear, guilt, shame, shyness, amusement, awe, contentment, gratitude, hope, love, pride, sympathy, and sexual feelings (e.g., "I felt sexual, desiring, and flirtatious"). The scale can be scored for total positive and negative affect,grouped according to where they would fall on the circumplex model of affect (e.g., high activation vs. lower activation),or individual affects can be examined. In student samples this modified DES has shown acceptable reliability with the positive affects subscale (α = .79) and the negative affects subscale (α = .69).

SECONDARY OUTCOMES:
Change in burden at end of intervention, 3 and 6-months post - Zarit Burden Inventory (Zarit, Reever, & Bach-Peterson, 1980) | Baseline and weeks 6 and 10; 3-months and 6-months post
  22-item inventory assesses caregivers' subjective feelings of the impact of caregiving on emotional and physical health functioning, social life, and financial status.
Change in perceived stress at end of intervention, 3 and 6-months post - Perceived Stress Scale (PSS) (Cohen, 1988) | Baseline and weeks 6 and 10; 3-months and 6-months post
  The 10 items are designed to identify how unpredictable, uncontrollable and overloaded respondents find their lives. Scores range from 0-40, with higher scores indicating greater stress.
Change in caregiver strain at end of intervention, 3 and 6-months post - Caregiver Strain Index (CSI) (Robinson, 1983) | Baseline and weeks 6 and 10; 3-months and 6-months post
  The CSI is a 13-item measure of both objective and subjective elements of caregiver strain.
Change in depression at end of intervention, 3 and 6-months post - Depression, Patient Reported Outcomes Measurement Information System Item Bank, v. 1.0 (PROMIS; Cella et al., 2010) | Baseline and weeks 6 and 10; 3-months and 6-months post
  Used to assess depressive mood.
Change in anxiety at end of intervention, 3 and 6-months post - Emotional Distress - Anxiety, PROMIS Item Bank v. 1.0 (Cella et al., 2010) | Baseline and weeks 6 and 10; 3-months and 6-months post
  Used to assess anxiety.
Change in coping at end of intervention, 3 and 6-months post - Ways of Coping Scale (Folkman, Lazarus, Pimley, & Novacek, 1987) | Baseline and weeks 6 and 10; 3-months and 6-months post
  The 23 forms of coping responses assessed include: confrontive coping, escape-avoidance, planful problem-solving, positive reappraisal, benefit, growth, mastery of stress, other success, purpose, positive relations with others, religion, and respite, benevolent and negative religious coping, emotional processing and expression, goal replacement, and maintaining optimism.

CONTACTS AND LOCATIONS:
Overall Officials: Glenna A Dowling, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Moskowitz JT, Cheung EO, Snowberg KE, Verstaen A, Merrilees J, Salsman JM, Dowling GA. Randomized controlled trial of a facilitated online positive emotion regulation intervention for dementia caregivers. Health Psychol. 2019 May;38(5):391-402. doi: 10.1037/hea0000680. PMID 31045422